CLINICAL TRIAL: NCT02324114
Title: Clinical Trial of Quantitative Detection Kit for Hsp90α in Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Protgen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: hsp90a2011-03
Record Dates: First submitted 2014-12-14; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Colorectal Cancer
Keywords: Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rectal cancer (Experimental): Detect plasma Hsp90α concentration of patients,
  Interventions: Device: Hsp90

INTERVENTIONS:
Device: Hsp90 — Detect plasma Hsp90α concentration
  Other Names: biomarker

SUMMARY:
Detect plasma Hsp90α concentration of colorectal cancer patients, healthy volunteers, benign colorectal diseases patients.

DETAILED DESCRIPTION:
Detect plasma Hsp90α concentration of colorectal cancer patients, healthy volunteers, benign colorectal diseases patients, validate accuracy, specificity and sensitivity of Hsp90α kit.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer patients, healthy volunteers, benign colorectal diseases patients

Exclusion Criteria:

* Patients who previously accepted radiotherapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Hsp90α Concentration(ng/ml) of plasma | 4 months
  Detect Hsp90α Concentration(ng/ml) of plasma and calculate the accuracy, specificity and sensitivity of Hsp90α kit

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, MD, Principal Investigator — Shandong province cancer hospital
Locations (1):
- Shandong province cancer hospital, Jinan, Shandong, China